CLINICAL TRIAL: NCT05212155
Title: Family-based Approach for Healthy Lifestyles (RYSE)
Brief Title: RYSE Family-based Behavioral Treatment for Childhood Obesity
Acronym: RYSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Children's Mercy Hospital Kansas City (Other); Freeman Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WU IRB 202103221
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Childhood
Keywords: behavioral treatment; lifestyle changes; exercise; Traffic Light Diet
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: The program is open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participating families (Other): Parent/child dyads enrolled in the open-label program
  Interventions: Behavioral: family-based behavioral treatment (FBT)

INTERVENTIONS:
Behavioral: family-based behavioral treatment (FBT) — Individual and group treatment of parent/child dyads to improve dietary choices, minimize sedentary behaviors, increase physical activity levels, and identify social support environments that reinforce healthy lifestyle choices.

SUMMARY:
RYSE is a Family-based Approach for Healthy Lifestyles that is a program for families with children between the ages of 5-12 years old to help them make healthy lifestyle changes to reach a healthier weight. The research program does this with children and their families through guidance about healthy eating, physical activity, and behavior change. The program focuses on helping participating families set up healthy support systems at home, at school and in social settings.

DETAILED DESCRIPTION:
Reducing the human and economic burden of obesity is a public health priority. Obesity disproportionately affects Black children (20% vs. 15% of White children)7 and low-income children. Family-based Behavioral Treatment (FBT) for childhood obesity is an effective, standardized behavioral intervention that has been developed and tested over the past 30 years by Drs. Leonard Epstein, Denise Wilfley, and colleagues. FBT targets both child and parent, with lasting positive effects that can extend to the family. FBT provides children and parents with new ways of thinking about their diet and exercise in order to support changes that support a healthy lifestyle. Participants work with "coaches" in individual sessions and in group sessions to both tailor the intervention to the family and provide an opportunity for social facilitation with other families that are participating. Missouri Medicaid (MOHealthNet) began reimbursement of 26 weeks of behavioral treatment for adult and child obesity on March 30, 2021. The FBT program implementation is designed to take advantage of this new benefit at clinical practices with the intent of creating a way to expand a workforce and standardize a program that can be disseminated across Missouri and possibly nationwide.

The purpose of the this research program is to evaluate for possible dissemination an online training program for FBT coaches, as well the implementation of the program, particularly in underserved rural and urban Black communities.

Participants comprise a dyad of parent and child. Full time caregivers that live with the dyad may participate in place of the parent, if the parent is unable to commit to the weekly sessions. Parental consent is required for the caregiver and the caregiver provides separate consent.

Participants attend weekly FBT group sessions with 3-10 participating families for 17 weeks, then 2 monthly individual sessions in month 5 and 6. This meets the 26-week Medicaid benefit requirement. Group sessions provide didactic content to support the families efforts to realign their diet and increase their exercise. Significant emphasis is placed on social networking, within the group session and in the participants' community, which is associated with better outcomes. There are 5 program sessions during the 6 months that are individual, with just the coach and the dyad. These are where program assessments are completed and the family and coach collaborate on goals and ways to meet them. The families also have two medical nutrition therapy consultations with registered dietitians. These are clinical interventions and not part of the research program structure. After the 26 weeks, the family returns for a 12-month research assessment, which is the final visit of the program.

When all participants have completed, matched-controls will be drawn from the electronic health record (EHR) at both clinical sites. Additional data are collected from the EHR to support cost analysis and implementation evaluation at the participant and organization levels.

This research program is being conducted at pediatric practices affiliated with Children's Mercy Hospital, Kansas City, MO and Freeman Health System, Joplin, MO. Washington University in St. Louis (WUSTL) is the primary award site and is responsible for FBT coach training and fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Parents ≥ 18 years old
* Children age 5-12 y, with BMI percentile ≥95th for age and sex
* Child must be enrolled in Missouri Medicaid
* Parent and child are comfortable speaking English
* Child is receiving primary care at one of the participating clinics
* Child lives with the participating parent ≥50% time
* Child able to provide written or verbal (based on age) informed assent,
* Child and parent able to participate in scheduled sessions

Exclusion Criteria:

* Parent/Caregiver is not the legal guardian of the child
* Purging (self-induced vomiting, diuretic use, laxative use) as an eating disorder
* Family lives ≥ 1 hour from the study sites
* Families planning to move out of the study area during the 12-month study period
* Child is a ward of the state

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Child weight change outcome | 25 weeks
  reduction, from baseline visit (BV), in child's percent overweight defined as (child's BMI - the median BMI [for the child's sex and age])/(median BMI) ×100

SECONDARY OUTCOMES:
Parent weight change outcome | 25 weeks
  percent change in weight from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Denise E Wilfley, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Freeman Health Pediatrics Clinics, Joplin, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Yes
All investigators on this project will be freely sharing data, with the PI collaborating with the co-investigators to coordinate the timing and topics of resulting publications.
  Access is restricted to de-identified data within 30 months following the end of data collection. Data requests may be sent in writing to the Principal Investigator, Denise Wilfley. Before being given access to the data, Protected Health Information (PHI) is removed and secondary users are asked to sign a data use agreement that defines conditions for the use of the data. Secondary users are asked to provide a brief description of the analyses they wish to perform. The restricted access agreement stipulates that the user is obliged to ensure the security and confidentiality of the data, that the data are used for Institutional Review Board (IRB)-approved purposes only, and that no effort will be made to identify individual participants.
Time Frame: 30 months after the database is closed.
Access Criteria: Coded dataset with IRB approval, limited dataset with HIPAA agreement, and de-identified dataset are accessible.